CLINICAL TRIAL: NCT07349069
Title: A Randomized, Open-Label, Phase III Trial to Compare HRS-8080 Versus Standard Endocrine Therapy in Patients With High-Risk Early Breast Cancer Who Have Received at Least 2 Years of Standard Adjuvant Endocrine Therapy
Brief Title: A Phase III Trial Comparing HRS-8080 With Standard Endocrine Therapy in Patients With High-Risk Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-305
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-8080 Group (Experimental): HRS-8080 tablets group.
  Interventions: Drug: HRS-8080 Tablets
- Letrozole or Tamoxifen Citrate Group (Active Comparator): Letrozole tablets or Tamoxifen Citrate tablets group.
  Interventions: Drug: Letrozole tablets; Drug: Tamoxifen Citrate Tablets

INTERVENTIONS:
Drug: HRS-8080 Tablets — HRS-8080 tablets.
  Arms: HRS-8080 Group
Drug: Letrozole tablets — Letrozole tablets.
  Arms: Letrozole or Tamoxifen Citrate Group
Drug: Tamoxifen Citrate Tablets — Tamoxifen Citrate tablets.
  Arms: Letrozole or Tamoxifen Citrate Group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-8080 in patients with high-risk early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 and ≤ 75 years with clinical stage II-III disease. Premenopausal patients must be willing to receive LHRH agonist therapy during the study period.
2. Histologically confirmed invasive breast cancer by postoperative pathology, having received at least 2 years, but no more than 5 years, of adjuvant endocrine therapy.
3. No evidence of recurrent or metastatic disease after surgery.
4. ECOG performance status of 0 or 1.
5. Adequate organ and bone marrow function.
6. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization and be willing to use acceptable non-hormonal contraception methods from the time of informed consent until 7 months after the last dose of the study drug.
7. Any acute toxicities from previous anti-tumor therapy have resolved to Grade 0-1 (per CTCAE v5.0).
8. The patient has provided written informed consent (ICF), and is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Tumor clinical stage IV (metastatic) breast cancer.
2. History and/or treatment of any malignancy other than breast cancer within 5 years prior to randomization.
3. History of severe pulmonary disease, such as interstitial lung disease.
4. Concurrent or potential use of any anti-tumor therapy not specified in the study protocol.
5. Major surgical procedure within 4 weeks prior to randomization.
6. HIV infection or known AIDS, active hepatitis B, hepatitis C, or co-infection with hepatitis B and C.
7. Poor cardiac function.
8. Severe infection within 4 weeks prior to randomization.
9. History of drug allergy.
10. History of organ transplantation.
11. History of substance abuse.
12. Women within 1 year postpartum or who are currently breastfeeding.
13. Patients deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
The time from the date of randomization to the first occurrence of any of the following events: ipsilateral local or contralateral invasive recurrence, distant recurrence, or death from any cause. | Every 26 weeks for the first 104 weeks after randomization, and then every 52 weeks thereafter, up to 5 years.
  Invasive Breast Cancer-Free Survival (IBCFS).

SECONDARY OUTCOMES:
Invasive Disease-Free Survival (IDFS). | Every 26 weeks for the first 104 weeks after randomization, and then every 52 weeks thereafter, up to 5 years.
Distant Metastasis-Free Survival (DRFS). | Every 26 weeks for the first 104 weeks after randomization, and then every 52 weeks thereafter, up to 5 years.
Overall Survival (OS). | Survival follow-up every 3 months, up to 5 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided